CLINICAL TRIAL: NCT03366298
Title: Pharmacokinetics of Intramuscular Adrenaline in Food--Allergic Teenagers: Does Dose Matter?
Brief Title: Pharmacokinetics of Intramuscular Adrenaline in Food--Allergic Teenagers
Acronym: PIMAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Paul Turner, MRC Clinician Scientist, Imperial College London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17SM4137; 2017-003239-13 (EudraCT Number); 232931 (Other: HRA)
Record Dates: First submitted 2017-11-21; First posted 2017-12-08 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Anaphylaxis
MeSH Terms: conditions — Anaphylaxis | interventions — Epinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 1 (Active Comparator): Visit 1: Emerade 300mcg then Epipen 0.3mg Visit 2: Emerade 500mcg
  Interventions: Combination Product: Epipen 0.3mg; Combination Product: Emerade 300mcg; Combination Product: Emerade 500mcg
- 2 (Active Comparator): Visit 1: Epipen 0.3mg then Emerade 300mcg Visit 2: Emerade 500mcg
  Interventions: Combination Product: Epipen 0.3mg; Combination Product: Emerade 300mcg; Combination Product: Emerade 500mcg
- 3 (Active Comparator): Visit 1: Emerade 500mcg Visit 2: Emerade 300mcg then Epipen 0.3mg
  Interventions: Combination Product: Epipen 0.3mg; Combination Product: Emerade 300mcg; Combination Product: Emerade 500mcg
- 4 (Active Comparator): Visit 1: Emerade 500mcg Visit 2: Epipen 0.3mg then Emerade 300mcg
  Interventions: Combination Product: Epipen 0.3mg; Combination Product: Emerade 300mcg; Combination Product: Emerade 500mcg

INTERVENTIONS:
Combination Product: Epipen 0.3mg — Epipen 0.3mg auto-injector
  Other Names: Epinephrine
Combination Product: Emerade 300mcg — Emerade 300mcg auto-injector
  Other Names: Epinephrine
Combination Product: Emerade 500mcg — Emerade 500mcg auto-injector
  Other Names: Epinephrine

SUMMARY:
Food allergy affects up to 2% of adults and 8% of children in the United Kingdom (UK), and is a major public health issue. It is the commonest cause of life-threatening allergic reactions (anaphylaxis), which can be fatal. Adrenaline (epinephrine) auto-injector (AAI) devices are the first-line treatment for anaphylaxis, yet in a UK survey, over 80% of 245 teenagers experiencing anaphylaxis did not use their AAI. Delays in, or lack of adrenaline (epinephrine) administration during anaphylaxis are risk factors for fatal anaphylaxis.

In 2010, a coroner's investigation into the death of a food-allergic teenager in the UK raised several questions around AAI safety and efficacy, since the teenager died despite administering her auto-injector device. This prompted a review by the Medicines and Healthcare products Regulatory Agency (MHRA) in 2014 into the clinical and quality considerations of AAIs. Two recommendations which came from the review was that companies 'should be encouraged to develop a 0.5mg [dose] AAI.' In the UK currently only Emerade, one of the three companies selling AAIs, manufactures a 0.5mg (500mcg) version. Emerade also has a longer needle length (23mm) compared to other AAIs (typically 15mm).

The investigators plan to formally assess the pharmacokinetics (PK) and pharmacodynamics (PD) of self-injection with intramuscular adrenaline (epinephrine) in teenagers at risk of anaphylaxis due to food allergy, and have been prescribed AAI.

1. The investigators will compare self-injection with 300mcg vs 500mcg in teenagers of body weight >40kg. In a 40kg person, an adrenaline dose of 300mcg results in an effective UNDER-dosing of 30% by body weight.
2. The investigators will also assess the impact of needle length on injection, by comparing two different devices, both of which deliver 300mcg, but one via a 15mm needle and the other with a 23mm needle.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 - 18 years inclusive
* Body mass >40kg
* Prescription of AAI due to physician diagnosis of Immunoglobulin E-mediated food allergy.
* Written informed consent from parent/guardian together with patient assent, for participants under 16 years of age. For young people age 16+ years, consent will be obtained from the participant themselves.

Exclusion Criteria:

* Known cardiac comorbidity (including hypertension, structural or electrophysiological diagnoses) or prescribed a medicine to control cardiovascular disease/hypertension.
* Known endocrine or renal disease
* Poorly controlled asthma requiring daily rescue treatment with a bronchodilator.
* Pregnancy
* Unwilling or unable to comply with study requirements

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, FRACP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London / Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Patel N, Isaacs E, Duca B, Nagaratnam N, Donovan J, Fontanella S, Turner PJ. Optimal dose of adrenaline auto-injector for children and young people at risk of anaphylaxis: A phase IV randomized controlled crossover study. Allergy. 2023 Jul;78(7):1997-2006. doi: 10.1111/all.15675. Epub 2023 Feb 23. PMID 36794963

RESULTS

PARTICIPANT FLOW:
Groups:
- Emerade 300 / Epipen 0.3mg / Emerade 500: Visit 1: Emerade 300mcg then Epipen 0.3mg Visit 2: Emerade 500mcg
  Epipen 0.3mg: Epipen 0.3mg auto-injector
  Emerade 300mcg: Emerade 300mcg auto-injector
  Emerade 500mcg: Emerade 500mcg auto-injector
- Epipen 0.3mg / Emerade 300 / Emerade 500: Visit 1: Epipen 0.3mg then Emerade 300mcg Visit 2: Emerade 500mcg
  Epipen 0.3mg: Epipen 0.3mg auto-injector
  Emerade 300mcg: Emerade 300mcg auto-injector
  Emerade 500mcg: Emerade 500mcg auto-injector
- Emerade 500 / Emerade 300 / Epipen 0.3mg: Visit 1: Emerade 500mcg Visit 2: Emerade 300mcg then Epipen 0.3mg
  Epipen 0.3mg: Epipen 0.3mg auto-injector
  Emerade 300mcg: Emerade 300mcg auto-injector
  Emerade 500mcg: Emerade 500mcg auto-injector
- Emerade 500 / Epipen 0.3mg / Emerade 300: Visit 1: Emerade 500mcg Visit 2: Epipen 0.3mg then Emerade 300mcg
  Epipen 0.3mg: Epipen 0.3mg auto-injector
  Emerade 300mcg: Emerade 300mcg auto-injector
  Emerade 500mcg: Emerade 500mcg auto-injector
Period: Overall Study
Arm/Group | Emerade 300 / Epipen 0.3mg / Emerade 500 | Epipen 0.3mg / Emerade 300 / Emerade 500 | Emerade 500 / Emerade 300 / Epipen 0.3mg | Emerade 500 / Epipen 0.3mg / Emerade 300
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Cohort: Overall study cohort
Arm/Group | Overall Cohort
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 15.4 [13.3 to 18.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Body Mass Index [Median (Full Range); unit: kg/m^2] | 20 [16.1 to 27.5]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Catecholamine Levels (Maximum Concentration, Cmax)
Description: Pharmacokinetics (plasma catecholamine levels: Cmax) following intramuscular self-injection of 300mcg and 500mcg adrenaline using an auto-injector device, in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Measure: Mean (95% Confidence Interval); unit: pg/ml
Groups:
- Emerade 300mcg Injection: Self-injection with Emerade 300mcg adrenaline auto-injector
- Emerade 500mcg Injection: Self-injection with Emerade 500mcg adrenaline auto-injector
- Epipen 0.3mg: Self-injection with Epipen 0.3mg adrenaline auto-injector
Arm/Group | Emerade 300mcg Injection | Emerade 500mcg Injection | Epipen 0.3mg
Number analyzed (Participants) | 12 | 12 | 12
pg/ml | 218 [132 to 359] | 394 [310 to 500] | 290 [200 to 421]

2. Primary Outcome: Plasma Catecholamine Levels (Time to Maximum Concentration, Tmax)
Description: Pharmacokinetics (plasma catecholamine levels: Tmax) following intramuscular self-injection of 300mcg and 500mcg adrenaline using an auto-injector device, in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Emerade 300mcg Injection | Emerade 500mcg Injection | Epipen 0.3mg
Number analyzed (Participants) | 12 | 12 | 12
minutes | 9.6 [5.3 to 17.4] | 8.5 [6.1 to 11.8] | 5.9 [4.9 to 7.3]

3. Primary Outcome: Plasma Catecholamine Levels (Maximum Concentration, Area-under-curve (AUC))
Description: Pharmacokinetics (plasma catecholamine levels: AUC) following intramuscular self-injection of 300mcg and 500mcg adrenaline using an auto-injector device, in food-allergic teenagers over 40kg.
  Baseline corrected.
Time Frame: At at the following timepoints following injection: 5, 10, 15, 20, 30, 45, 60, 80, 100, 120 and 180 minutes
Measure: Mean (95% Confidence Interval); unit: hr*pg/ml
Arm/Group | Emerade 300mcg Injection | Emerade 500mcg Injection | Epipen 0.3mg
Number analyzed (Participants) | 12 | 12 | 12
hr*pg/ml | 174 [86 to 354] | 387 [263 to 570] | 203 [142 to 292]

4. Secondary Outcome: Change in Heart Rate Following Self-injection of Adrenaline (300mcg, 500mcg) on Separate Occasions.
Description: Pharmacodynamics (heart rate) following intramuscular self-injection of 300mcg and 500mcg adrenaline using an auto-injector device, in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

5. Secondary Outcome: Change in Blood Pressure Following Self-injection of Adrenaline (300mcg, 500mcg) on Separate Occasions.
Description: Pharmacodynamics (blood pressure) following intramuscular self-injection of 300mcg and 500mcg adrenaline using an auto-injector device, in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

6. Secondary Outcome: Change in Stroke Volume Following Self-injection of Adrenaline (300mcg, 500mcg) on Separate Occasions.
Description: Pharmacodynamics (stroke volume) following intramuscular self-injection of 300mcg and 500mcg adrenaline using an auto-injector device, in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

7. Secondary Outcome: Impact of Needle Length on Pharmacokinetics (Plasma Catecholamine Levels: Cmax)
Description: Pharmacokinetics (plasma catecholamine levels: Cmax) following intramuscular self-injection of 300mcg adrenaline using two auto-injector devices with different needle lengths (15mm vs 23mm), in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

8. Secondary Outcome: Impact of Needle Length on Pharmacokinetics (Plasma Catecholamine Levels: Tmax)
Description: Pharmacokinetics (plasma catecholamine levels: Tmax) following intramuscular self-injection of 300mcg adrenaline using two auto-injector devices with different needle lengths (15mm vs 23mm), in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

9. Secondary Outcome: Impact of Needle Length on Pharmacokinetics (Plasma Catecholamine Levels: AUC)
Description: Pharmacokinetics (plasma catecholamine levels: AUC) following intramuscular self-injection of 300mcg adrenaline using two auto-injector devices with different needle lengths (15mm vs 23mm), in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

10. Secondary Outcome: Impact of Needle Length on Pharmacodynamics (Cardiovascular Parameters: Heart Rate)
Description: The pharmacodynamics (cardiovascular parameters: heart rate) following intramuscular self-injection of 300mcg adrenaline using two auto-injector devices with different needle lengths (15mm vs 23mm), in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

11. Secondary Outcome: Impact of Needle Length on Pharmacodynamics (Cardiovascular Parameters: Blood Pressure)
Description: The pharmacodynamics (cardiovascular parameters: blood pressure) following intramuscular self-injection of 300mcg adrenaline using two auto-injector devices with different needle lengths (15mm vs 23mm), in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

12. Secondary Outcome: Impact of Needle Length on Pharmacodynamics (Cardiovascular Parameters: Stroke Volume)
Description: The pharmacodynamics (cardiovascular parameters: stroke volume) following intramuscular self-injection of 300mcg adrenaline using two auto-injector devices with different needle lengths (15mm vs 23mm), in food-allergic teenagers over 40kg.
Time Frame: 3 hours
Reporting Status: Not Posted

13. Secondary Outcome: Adverse Events Following Self-administration of Adrenaline Via Autoinjector Device
Description: Adverse events following self-administration of adrenaline via autoinjector device defined as in protocol
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Emerade 300mcg Injection | Emerade 500mcg Injection | Epipen 0.3mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Pain at injection site | 8 | 6 | 7
  Systemic AE (any) | 4 | 9 | 8
  Palpitations | 3 | 4 | 3
  Tremor | 3 | 7 | 8

14. Secondary Outcome: Change in Health-related Quality of Life (HRQL) as Measured Using FAQLQ
Description: The impact of self-administration of adrenaline autoinjectors (in a non-reaction setting) on health-related quality of life (HRQL) measures in food-allergic teenagers and their parents.
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Within 24h of injection only
Arm/Group | Emerade 300mcg Injection | Emerade 500mcg Injection | Epipen 0.3mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 9/12 | 8/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Emerade 300mcg Injection (N=12) | Emerade 500mcg Injection (N=12) | Epipen 0.3mg (N=12)
Palpitations (Cardiac disorders) | 3 (3) | 4 (4) | 3 (3)
Tremor (Nervous system disorders) | 3 (3) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT03366298/Prot_SAP_000.pdf